CLINICAL TRIAL: NCT05207891
Title: Comparing Two Types of Dynamic Air Mattresses, With Focus on Changes in Pressure Injury Occurrence and Functionality
Brief Title: Comparing Pressure Injury Occurrence in Patients Using Two Different Mattresses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sunnaas Rehabilitation Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: Mattress Comparison
Record Dates: First submitted 2021-09-27; First posted 2022-01-26 (Actual); Last update posted 2023-04-14 (Actual); Status verified 2023-04

CONDITIONS: Pressure Injury; Sleep; Pain; Satisfaction, Patient; Noise Exposure; Strains; Satisfaction, Personal
MeSH Terms: conditions — Pressure Ulcer; Pain; Patient Satisfaction; Sprains and Strains; Personal Satisfaction

STUDY DESIGN:
Intervention Model Description: Inclusion, collection of baseline data at day zero, then seven days use of the first mattress and data collection on day seven, new pressure measurement at day seven, seven days use of the second mattress and final data collection after seven days of use of the second mattress. Summarized, the data collection will be at baseline, at day seven and at day 14.
Masking Description: No masking. This will be an open label study, because it will be impossible to mask the mattresses due to different lay-out and function.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention mattress (Experimental): At every shift during the seven days project period, the nurses will check for pressure wounds, and mark identified pressure wounds and their category on a pressure injury body map. At every shift the nurses will use a custom made form to register resources needed in each position changing of the patient, the number of times the position is changed, as well as the level of physical strain in the nurses. All participants will start with seven days use of the newly developed intervention mattress. At the end of the testing period, the participants will register their feeling of quality of life, bedrest comfort, sleep-wellness, pain and satisfaction in the study period.
  A custom made semi-structured interview guide has been conducted asking in more details of experienced quality in use and in managing the mattress. One participant and one nurse will be asked to participate in in-depth interviews after testing both mattresses.
  Interventions: Device: Intervention mattress
- Regulare care mattress (No Intervention): At every shift during the seven days project period, the nurses will check for pressure wounds, and mark identified pressure wounds and their category on a pressure injury body map. At every shift the nurses will use a custom made form to register resources needed in each position changing of the patient, the number of times the position is changed, as well as physical strain in the nurses. At the end of the testing period, the participants will register their feeling of quality of life, bedrest comfort, sleep-wellness, pain and satisfaction in the test period.
  A custom made semi-structured interview guide has been conducted asking in more details of experienced quality in use and in managing the mattress. One participant and one nurse will be asked to participate in in-depth interviews after testing both mattresses.

INTERVENTIONS:
Device: Intervention mattress — The intervention mattress, Tidewave, will be compared to the regular care mattress, CuroCell 4AD. Primary outcome will be change in pressure injury occurence, assessed according to the NPIAP 2019 Clinical Guidance, and marked up on pressure injury body-map figures. Secondary outcomes will be experienced quality of life, assessed with the Spinal Cord Injury Quality of Life Basic Data Set. Further mattress comfort, assessed with the Mattress Comfort Scale, sleep-wellness, assessed with the Insomnia Severity Index, and pain, assessed with the Brief Pain Inventory. Satisfaction in the participants and in the nursing staff will be assessed with custom made Likert scales. Resource use and experienced stain in the nursing staff will be assessed with custom made forms asking for number of persons needed in position change, number of position changes needed during bed-rest, and experienced strain related to the position changes.
  Other Names: Tidewave
  Arms: Intervention mattress

SUMMARY:
The purpose of this project is to compare a newly developed automatic reversing dynamic air mattress, with a regular care mattress, which is in daily use at the hospital. Focus will be on pressure relief in relation to occurrence of pressure injury, user satisfaction, and the mattresses impact on sleep and pain. The participants will be randomized to start with the intervention mattress or the control mattress. Outcomes will be measured via validated forms regarding pressure related injuries, quality of life, pain, and mattress comfort. Custom made forms will be used regarding resource use and comfort in the nursing service, especially in relation to position changes in the participants .

DETAILED DESCRIPTION:
The investigators will conduct a randomized cross over testing, where the purpose is to compare an intervention mattress and a regular care mattress in relation to occurrence of pressure relief, experienced sleep comfort, pain and quality of life in the participants. Further on, the investigators want to examine staff needed to assist in position change of the participants, as well as physical strain for the staff.

To secure safe use of the intervention mattress, a noise-test and a pressure assessment test of the mattresses have been performed in advance of the research project. A pressure limit is defined, based on current evidence based knowledge regarding pressure injury risk. If this limit is exceeded during the project period, the participant will be excluded from further testing, due to a potential increased risk of pressure injury development.

Written and oral information regarding the project will be given, and the participants will give a written concent before inclusion.

The regular care mattress, used as control in this trial, is considered one of the best pressure relieving mattresses available in Norway.

Ten participants will be included and randomized to start with the intervention mattress or the control mattress. Baseline data regarding gender, age, level and severity of the spinal injury, together with pressure injury associated dysfunction, like increased sweat, bladder and bowel incontinency will be collected immediately after inclusion. The investigators will also ask for information of comorbidity previous to the spinal injury, including cardiovascular disease, embolisms or diabetes mellitus.

Pressure monitoring will be performed before start up, and validated questionnaires will be used in assessing pressure injury risk, pain and quality of life. Pressure injury occurrence will be assessed every day. After seven days use of the first mattress, new data will be collected, by means of validated forms regarding pain occurrence, noise from the mattress devices, sleeping wellness and participant satisfaction. Custom made forms regarding resource use in the nursing staff, especially at night and in relation to position change, will be collected, together with data regarding physical strain in the staff.

The participant will then change to the other mattress and pressure monitoring will be performed. If acceptable results, the participant will use this mattress for seven days. Pressure injury occurrence will be assessed every day. Then a end-of-study data assessment will be performed, similar to the questionnaires used in the intervention mattress.

Finally, in-depth interviews will be performed in one participants and one nurse finishing the study on the intervention mattress, and one participant and one nurse finishing the study, using the control mattress.

ELIGIBILITY:
Inclusion Criteria:

* > 18 years of age
* SCI, neurological disease with paralysis or multi trauma, all with lack of independency in position change in bed, and hospitalized for primary rehabilitation in either the Spinal Cord Unit (SCU) or the Multi trauma, Neurological disease, Burn (MNB) Unit
* Requires manual position change
* Medically approved for the participation by the participant's physician
* Able to give consent to participate
* Psychically and cognitively able to properly answer the questionnaires
* Speaks/understands Norwegian language

Exclusion Criteria:

* Ongoing pressure injury
* External fixation, except neck collar
* Body weight > 150 kg
* pre-test pressure assessment above the maximum pressure limit.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2021-09-14 (Actual); Primary Completion 2023-03-01 (Actual); Study Completion 2023-03-01 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in the pressure injury risk will be assessed via the Braden Scale at study completion at day 14. | Pressure injury risk assessment will be performed at baseline (day zero) and at study completion at day 14.
  The Braden scale assesses a patient's risk of developing a pressure injury by examining the patient's sensory perception related to discomfort or pain caused by pressure. Further, the scale assesses the degree of moisture the skin is exposed to, level of physical activity, the capability and willingness of a patient to adjust the body positioning independently, the nutritional status and the amount of assistance a patient needs to move, as well as the degree of sliding in bed or chair. The total rating of each of these categories gives an indication of the pressure injury risk for the specific person.
Change in pressure injury occurence from (day zero), will be assessed, via the National Pressure Injury Advisory Panel 2019 Guideline, once a day to study completion at day 14. | Pressure injury occurence will be assessed from baseline (day zero) and once a day to study completion at day 14.
  Pressure injury assessment will be performed with categorization of any occuring pressure injuries in accordance with the National Pressure Injury Advisory Panel 2019 Guideline, regarding severity of the pressure injury.

SECONDARY OUTCOMES:
Change in Quality of Life (QoL) from baseline, will be assessed via the spinal cord injury quality of Life basic data set (SCI QoL BDS) at day seven, and at day conclusion of the study at day 14. | Assessment will be performed at baseline (day zero), at change of mattress at day seven, and at study conclusion, at day 14.
  Self-assessment will be performed, using the spinal cord injury quality of life basic data set (SCI QoL BDS), with a Likert scale from 0 to 10, where all numbers, including 0 can be used, and where 10 is the best possible health, while 0 is the worst possible.
Change from baseline in the sleep wellness will be assessed via the Insomnia Severity Index (ISI) at day seven and at conclusion of the study at day 14. | Assessment will be performed at baseline (day zero), at change of mattress at day seven, and at study completion at day 14.
  Assess the sleep wellness for the past 7 days, using the Insomnia Severity Index (ISI), consisting of seven questions, each with five possible answers going from no problem (0 points) to severe problem (4 points). The seven answers will then be added up, and the total score gives a numeric indication of the sleep wellness, with 0 to 7 points indicating absence of insomnia, 8 to 14 indicating sub-threshold insomnia, 15 to 21 indicating moderate insomnia, and 22 to 28 indicating severe insomnia.
Change in participant satisfaction from baseline, will be assessed via a custom made Likert scale at day seven, and at conclusion of the study at day 14. | Assessment will be performed at baseline (day zero), at change of mattress at day seven, and at study completion at day 14.
  Assess the participant satisfaction using the mattresses, via a custom made Likert scale, where 1 is completely dissatisfied, and 5 is totally satisfied.
Change in staff satisfaction from baseline, will be assessed via a custom made Likert scale at day seven, and at conclusion of the study at day 14. | Assessment will be performed at baseline (day zero), at change of mattress at day seven, and at study completion at day 14.
  Assess the staff's satisfaction with the mattress regarding body strain. The assessment will be performed via a custom made Likert scale, where 1 is completely dissatisfied, and 5 is totally satisfied.
Change in pain intensity from baseline will be assessed via the Brief Pain Inventory (BPI) form at change of mattress at day seven, and at end of study at day 14. | Assessment will be performed at baseline (day zero), at change of mattress at day seven, and at study completion at day 14.
  Assess experienced pain, using the the pain intensity part of the Brief Pain Inventory (BPI). The participants will perform a self-assessment of the pain intensity, they experience at the time of assessment, on a 0 to 10 scale where 0 being no pain and 10 being the worst possible pain.
Change in pain's interference with functions from baseline will be assessed via the Brief Pain Inventory form at day seven and at day 14. | Assessment will be performed at baseline (day zero), at change of mattress at day seven, and at study completion at day 14.
  The interference part of the Brief Pain Inventory (BPI) form will be used. The participants will perform a self-assessment of their pain's interference with functions, regarding general activity, walking, work, mood, enjoyment of life, relations with others, and sleep. Each of the activities will be scored on a 0 to 10 scale, where 0 being no interference at all, and 10 being the worst possible interference.The pain interference will be scored as the mean of the seven activities assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Ingebjørg Irgens, MD, Principal Investigator — Sunnaas Rehabilitation Hospital
Locations (1):
- Sunnaas Rehabilitation Hospital, Nesoddtangen, Akershus, Norway

IPD SHARING:
Plan to Share IPD: Yes
Data from the pressure measurement and questionnaires will be shared.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Time for sharing is planned to open in 2024, after finishing the study and analysing the data.
Access Criteria: On request, and in accordance with the Norwegian privacy protecting legislation

DOCUMENTS (2):
  • Study Protocol (2022-01-01): https://cdn.clinicaltrials.gov/large-docs/91/NCT05207891/Prot_000.pdf
  • Informed Consent Form (2022-01-01): https://cdn.clinicaltrials.gov/large-docs/91/NCT05207891/ICF_001.pdf